CLINICAL TRIAL: NCT03086265
Title: The Safety and Efficacy of the Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) for Laser Laryngeal Surgery
Brief Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) and Laser Laryngeal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vladimir Nekhendzy, Clinical Professor of Anesthesiology and Otolaryngology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36060
Record Dates: First submitted 2017-03-05; First posted 2017-03-22 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Otorhinolaryngologic Surgical Procedures; Laser Therapy
Keywords: airway management; high flow nasal oxygen high flow nasal cannula THRIVE; high flow nasal cannula THRIVE; THRIVE
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- THRIVE (Experimental): high flow nasal oxygen
  Interventions: Device: THRIVE
- Endotracheal tube (Active Comparator): tracheal intubation
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: THRIVE — active nasal oxygen delivery system
  Arms: THRIVE
Device: Endotracheal tube — Plastic tube for supporting ventilation during surgery
  Arms: Endotracheal tube

SUMMARY:
The purpose of this study is to investigate whether laser laryngeal surgery can be safely and potentially more effectively performed without the use of tracheal intubation or jet ventilation, under completely tubeless conditions. The patient's gas exchange will be supported by rapid insufflation of high-flow oxygen through specialized nasal cannula: the so called Transnasal Humidified Rapid- Insufflation Ventilatory Exchange (THRIVE).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for laser laryngeal surgery

Exclusion Criteria:

1. Patients with significantly decreased myocardial function (ejection fraction < 50%)
2. Patients with abnormal cardiac rhythm and conduction abnormalities, except for patients with isolated, asymptomatic premature atrial and ventricular contractions.
3. Patients with significant peripheral vascular disease, such as those with the symptoms of intermittent claudication.
4. Patients with known significant cerebrovascular disease, such as history of cerebrovascular accidents (CVAs) and transient ischemic attacks (TIAs) .
5. Patients with significant renal insufficiency, as manifested by estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2.
6. Patients with electrolyte (K+, Ca++) abnormalities, as determined by the lab values outside of a normal range.
7. Patients with the history or symptoms of increased intracranial pressure or reduced intracranial compliance (e.g. headaches, nausea and vomiting, visual changes, mental changes).
8. Patients with skull base defects.
9. Patients with pulmonary hypertension who have pulmonary artery pressures above the normal range.
10. Patients with significant chronic obstructive or restrictive lung diseases, as manifested by known history of baseline chronic hypoxia and/or hypercapnia, and/or baseline room air oxygen saturation (SpO2) < 95% .
11. Obese patients with BMI > 35 kg/m2.
12. Patients with severe and poorly controlled gastroesophageal reflux disease despite medical treatment.
13. Patients with hiatal hernia and full stomach patients.
14. Patient's refusal to participate in the study.
15. Patients who do not understand English or mentally handicapped. Pregnant or breastfeeding patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Nekhendzy, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- THRIVE: Participants received high flow nasal oxygen (THRIVE: active nasal oxygen delivery system).
- Endotracheal Tube: Participants received tracheal intubation (endotracheal tube: Plastic tube for supporting ventilation during surgery).
Period: Overall Study
Arm/Group | THRIVE | Endotracheal Tube
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THRIVE | Endotracheal Tube | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15) | 52 (12) | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Lowest Intraoperative Peripheral Oxygen Saturation (SpO2)
Description: Peripheral oxygen saturation is an estimate of the amount of oxygen in the blood.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
percentage of oxygen | 97 (2) | 97 (3)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.7934, t-test, 2 sided

2. Primary Outcome: Partial Pressure of Oxygen in the Arterial Blood (PaO2)
Time Frame: Induction, 10, 20, 30, 40m following induction, spontaneous ventilation (approximately 1 hour), recovery room (approximately 1 hour)
Population: This outcome was assessed in THRIVE participants only. Participants with measurements at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | THRIVE
Number analyzed (Participants) | 10
mmHg
  Induction | 365 (40)
  10 minutes post-induction | 294 (79)
  20 minutes post-induction | 279 (81)
  30 minutes post-induction | 245 (81)
  40 minutes post-induction: number analyzed (Participants) | 6
  40 minutes post-induction | 223 (67)
  Spontaneous ventilation | 251 (102)
  Recovery room | 86 (13)

3. Primary Outcome: Partial Pressure of Carbon Dioxide in the Arterial Blood (PaCO2)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | THRIVE
Number analyzed (Participants) | 10
mmHg
  Induction | 32 (5)
  10 minutes post-induction | 54 (5)
  20 minutes post-induction | 65 (9)
  30 minutes post-induction | 77 (8)
  40 minutes post-induction: number analyzed (Participants) | 6
  40 minutes post-induction | 86 (7)
  Spontaneous ventilation | 71 (13)
  Recovery room | 37 (5)

4. Primary Outcome: pH in Blood
Description: The pH range is 0 to 14, with 7 being neutral. A pH of less than 7 indicate acidity, whereas a pH of greater than 7 indicates a base.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | THRIVE
Number analyzed (Participants) | 10
pH
  Induction | 7.4 (0)
  10 minutes post-induction | 7.2 (0)
  20 minutes post-induction | 7.2 (0)
  30 minutes post-induction | 7.1 (0)
  40 minutes post-induction: number analyzed (Participants) | 6
  40 minutes post-induction | 7.1 (0.1)
  Spontaneous ventilation | 7.4 (0.1)
  Recovery room | 7.4 (0)

5. Primary Outcome: Heart Rate
Time Frame: Induction, 10, 20, 30, 40m following induction, spontaneous ventilation (approximately 1 hour)
Population: Participants with measurements at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
beats per minute
  Induction | 65 (11) | 70 (15)
  10 minutes post-induction | 72 (12) | 81 (14)
  20 minutes post-induction | 79 (13) | 79 (9)
  30 minutes post-induction | 79 (14) | 76 (12)
  40 minutes post-induction: number analyzed (Participants) | 6 | 10
  40 minutes post-induction | 81 (15) | 73 (9)
  Spontaneous ventilation | 72 (14) | 71 (15)

6. Primary Outcome: Mean Arterial Pressure (MAP)
Time Frame: Induction, 10, 20, 30, 40m following induction, spontaneous ventilation (approximately 1 hour)
Population: Participants with measurements at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
mmHg
  Induction | 90 (16) | 92 (12)
  10 minutes post-induction | 78 (12) | 76 (9)
  20 minutes post-induction | 71 (9) | 83 (17)
  30 minutes post-induction | 72 (12) | 85 (13)
  40 minutes post-induction: number analyzed (Participants) | 6 | 10
  40 minutes post-induction | 69 (13) | 80 (12)
  Spontaneous ventilation | 88 (14) | 88 (18)

7. Primary Outcome: Stroke Volume Index (SVI)
Description: Stroke volume - the volume of blood ejected from a ventricle at each beat of the heart, equal to the difference between the end-diastolic volume and the end-systolic volume. The stroke volume index is a method of relating the stroke volume to the size of the person by dividing the stroke volume by the body surface area (BSA) (m^2).
Time Frame: Induction, 10, 20, 30, 40m following induction, spontaneous ventilation (approximately 1 hour)
Population: Participants with measurements at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: ml/b/m^2
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
ml/b/m^2
  Induction | 50 (10) | 48 (13)
  10 minutes post-induction | 45 (7) | 36 (7)
  20 minutes post-induction | 48 (10) | 35 (6)
  30 minutes post-induction | 51 (12) | 39 (9)
  40 minutes post-induction: number analyzed (Participants) | 6 | 10
  40 minutes post-induction | 52 (6) | 43 (10)
  Spontaneous ventilation | 54 (17) | 53 (12)

8. Primary Outcome: Cardiac Index (CI)
Description: Cardiac index: A cardiodynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area (m^2) to yield the cardiac index.
Time Frame: Induction, 10, 20, 30, 40m following induction, spontaneous ventilation (approximately 1 hour)
Population: Participants with measurements at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
L/min/m^2
  Induction | 3.2 (0.7) | 3.4 (0.9)
  10 minutes post-induction | 3.2 (0.7) | 3.0 (0.7)
  20 minutes post-induction | 3.7 (0.5) | 2.8 (0.5)
  30 minutes post-induction | 3.9 (0.7) | 3.0 (0.6)
  40 minutes post-induction: number analyzed (Participants) | 6 | 10
  40 minutes post-induction | 4.2 (0.8) | 3.1 (0.7)
  Spontaneous ventilation | 3.7 (0.9) | 3.6 (0.6)

9. Primary Outcome: Systemic Vascular Resistance Index (SVRI)
Description: SVRI equals systemic vascular resistance (SVR) times BSA. SVR is the resistance to blood flow through the systemic circulation and it was measured in Wood units. Wood unit =80 dyne*seconds per centimetre^5 (dyne*sec/cm^5).
Time Frame: Induction, 10, 20, 30, 40m following induction, spontaneous ventilation (approximately 1 hour)
Population: Participants with measurements at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: dynes*s/cm^5/m^2
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
dynes*s/cm^5/m^2
  Induction | 2249 (652) | 2140 (443)
  10 minutes post-induction | 1769 (549) | 2026 (446)
  20 minutes post-induction | 1341 (321) | 2182 (440)
  30 minutes post-induction | 1330 (464) | 2080 (446)
  40 minutes post-induction: number analyzed (Participants) | 6 | 10
  40 minutes post-induction | 1130 (217) | 1187 (530)
  Spontaneous ventilation | 1841 (443) | 2152 (578)

10. Primary Outcome: Awakening/Extubation Time
Description: Recorded from the end of surgery until the return of patient's protective airway reflexes and patient opening eyes to command.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 14 (3) | 13 (6)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.6876, t-test, 2 sided

11. Primary Outcome: Time to Suspension
Description: Recorded from the moment of the introduction of the operating laryngoscope in patient's mouth to full surgical suspension.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 4 (2) | 3 (2)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.7549, t-test, 2 sided

12. Primary Outcome: Number of Suspension Adjustments
Description: Number of adjustments of the suspension laryngoscope.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: adjustments
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
adjustments | 1 (1) | 2 (4)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.6479, t-test, 2 sided

13. Primary Outcome: Duration of Surgery
Description: Recorded from the moment of the introduction of the operating laryngoscope in patient's mouth to withdrawing the laryngoscope at the completion of surgery.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 61 (29) | 57 (44)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.8322, t-test, 2 sided

14. Secondary Outcome: Count of Participants Requiring Jet Ventilation
Description: Jet ventilation refers to delivery of oxygen via high pressure jet ventilator.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
Participants | 7 | 0

15. Secondary Outcome: Time to Spontaneous Ventilation
Description: Recorded from the discontinuation of anesthetic drugs to the return of patient's spontaneous ventilation.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 5 (4) | 11 (5)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.0058, t-test, 2 sided

16. Secondary Outcome: Apnea Time
Description: Recorded from induction of anesthesia to the return of spontaneous ventilation.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 70 (28) | 87 (48)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.3346, t-test, 2 sided

17. Secondary Outcome: Duration of Anesthesia
Description: Recorded from induction of anesthesia to patient's awakening/extubation
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 78 (28) | 89 (48)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.5513, t-test, 2 sided

18. Secondary Outcome: Total Propofol Dose (Anesthetic)
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
mg | 730 (288) | 920 (388)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.1927, t-test, 2 sided

19. Secondary Outcome: Total Remifentanil Dose (Anesthetic)
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
µg | 996 (674) | 1114 (432)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.6483, t-test, 2 sided

20. Secondary Outcome: Total Phenylephrine Dose (Vasoactive Drug)
Time Frame: Duration of surgery (average approximately 1 hour)
Population: Participants who received phenylephrine are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 6 | 4
mg | 300 (591) | 479 (757)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.5625, t-test, 2 sided

21. Secondary Outcome: Total Ephedrine Dose (Vasoactive Drug)
Time Frame: Duration of surgery (average approximately 1 hour)
Population: Participants who received ephedrine are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 3 | 2
mg | 4 (8) | 1 (2)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.2827, t-test, 2 sided

22. Secondary Outcome: Total Labetalol Dose (Vasoactive Drug)
Time Frame: Duration of surgery (average approximately 1 hour)
Population: Participants who received labetalol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 3 | 6
mg | 15 (22) | 13 (21)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.8426, t-test, 2 sided

23. Secondary Outcome: Time to Patient Being Alert and Oriented x 4
Description: Recorded from patient's admission to the recovery room to patient's orientation to person, place, time, and situation as assessed by the recovery room nurse.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 23 (29) | 23 (19)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.9856, t-test, 2 sided

24. Secondary Outcome: Recovery Room Discharge-ready Time
Description: From admission to recovery room, to discharge from recovery room
Time Frame: Duration of recovery room stay (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
minutes | 64 (18) | 62 (12)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.8112, t-test, 2 sided

25. Secondary Outcome: First Pain Score in Recovery Room
Description: Pain scale was 0-10 (0 = no pain, 10 - worst pain imaginable).
Time Frame: Duration of recovery room stay (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
score on a scale | 2 (4) | 3 (3)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.6587, t-test, 2 sided

26. Secondary Outcome: Pain Score at Discharge From Recovery Room
Description: Pain scale was 0-10 (0 = no pain, 10 - worst pain imaginable).
Time Frame: Duration of recovery room stay (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
score on a scale | 3 (2) | 2 (2)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.4143, t-test, 2 sided

27. Secondary Outcome: Analgesic Consumption
Description: Analgesic consumption was measured in oral morphine milligram equivalents (MME)
Time Frame: Recovery room to 7th postoperative day
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
MME | 12 (17) | 8 (7)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Test type: Other; p = 0.4324, t-test, 2 sided

28. Secondary Outcome: Quality of Recovery (QoR)15 Score
Description: The QoR15 has 15 questions each is on a scale of 0-10 to measure patient functionality. Scores are summed for an overall range of 0-150, with higher scores corresponding to better recovery.
Time Frame: Prior to procedure, and 1-2 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Endotracheal Tube
Number analyzed (Participants) | 10 | 10
score on a scale
  Preoperative | 135 (17) | 138 (8)
  Postoperative | 146 (5) | 136 (11)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube; Comparison of preoperative scores; Test type: Other; p = 0.7221, t-test, 2 sided
Statistical Analysis 2: Comparison: THRIVE vs Endotracheal Tube; Comparison of postoperative scores; Test type: Other; p = 0.0336, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 1 week
Arm/Group | THRIVE | Endotracheal Tube
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03086265/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT03086265/SAP_001.pdf